CLINICAL TRIAL: NCT03591484
Title: Treatment of Halitosis With Photodynamic Therapy in Older Patients: Protocol for a Randomized, Controlled Trial
Brief Title: Treatment of Halitosis With Photodynamic Therapy in Older Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Halidosos
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2018-07

CONDITIONS: Halitosis
Keywords: Halitosis; photodynamic therapy; bronchiectasis
MeSH Terms: conditions — Halitosis; Bronchiectasis | interventions — Photochemotherapy; Therapeutics; Periodontal Index; Dentures

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G1 dentate healthy older (Experimental): Treatment with Photodynamic therapy (n = 20). The dentate participants will received periodontal treatment. The evaluation of halitosis and the microbiological analysis will be repeated before these steps
  Interventions: Radiation: Photodynamic therapy; Procedure: Periodontal treatment
- G2 healthy older/dentures (Experimental): Treatment with Photodynamic therapy (n = 20). The participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis and the microbiological analysis will be repeated before these steps
  Interventions: Radiation: Photodynamic therapy; Procedure: hygiene procedures for the mucosa and dentures
- G3 dentate older bronchiectasis (Active Comparator): Treatment with tongue scraper (n = 20). The dentate participants with bronchiectasis will received periodontal treatment. The evaluation of halitosis and the microbiological analysis will be repeated before these steps
  Interventions: Device: Treatment with tongue scraper; Procedure: Periodontal treatment
- G4 older bronchiectasis /dentures (Active Comparator): Treatment with tongue scraper (n = 20). The participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis and the microbiological analysis will be repeated before these steps
  Interventions: Device: Treatment with tongue scraper; Procedure: hygiene procedures for the mucosa and dentures

INTERVENTIONS:
Radiation: Photodynamic therapy — Treatment with Photodynamic therapy. The evaluation of halitosis and the microbiological analysis will be repeated before this step
  Arms: G1 dentate healthy older; G2 healthy older/dentures
Device: Treatment with tongue scraper — Treatment with tongue scraper. The evaluation of halitosis and the microbiological analysis will be repeated before this step
  Arms: G3 dentate older bronchiectasis; G4 older bronchiectasis /dentures
Procedure: Periodontal treatment — Periodontal treatment will be performed with curettes and ultrassom. The evaluation of halitosis and the microbiological analysis will be repeated before this step
  Arms: G1 dentate healthy older; G3 dentate older bronchiectasis
Procedure: hygiene procedures for the mucosa and dentures — edentulous participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis and the microbiological analysis will be repeated before this step
  Arms: G2 healthy older/dentures; G4 older bronchiectasis /dentures

SUMMARY:
Halitosis is the term used to define an unpleasant odor emanating from the mouth. Some lung diseases, such as bronchiectasis, are among the extra-oral causes of this condition. However, no studies have evaluated the causes and treatment of halitosis in the population of older adults with bronchiectasis. Methods and analysis: A randomized, controlled trial is proposed. The patients will be divided into four groups: G1- healthy older adults with 10 teeth or more (n = 40); G2- healthy older adults who wear complete dentures (n = 40); G3- older adults with bronchiectasis and 10 teeth or more (n = 40); and G4- older adults with bronchiectasis who wear complete dentures (n = 40). Halitosis will be evaluated based on the measurement of volatile sulfur compounds using gas chromatography. The participants with halitosis will be randomized into two subgroups: treatment with photodynamic therapy (n = 20) or cleaning of the tongue with a tongue scraper (n = 20). After the treatments, a second evaluation will be performed, along with a microbiological analysis (qPCR) for the identification of the bacteria P. gingivalis and T. denticola. If the halitosis persists, the dentate participants will received periodontal treatment and the edentulous participants will be submitted to hygiene procedures for the mucosa and dentures. The evaluation of halitosis and the microbiological analysis will be repeated. If the halitosis is resolved, the participants will return after three months for an additional evaluation. This protocol will determine the effectiveness of phototherapy regarding the reduction of halitosis in healthy older adults and those with bronchiectasis.

DETAILED DESCRIPTION:
Methods:

A single-center, randomized, controlled, single-blind clinical trial was designed in accordance with the criteria recommended for interventional trials in the SPIRIT Statement. The project for the proposed study received approval from the Human Research Ethics Committee of Universidade Nove de Julho (certificate number: 87160418.7.0000.5511).

Selection of individuals - characterization of sample - One group will be composed of older adults (60 years or older) with a diagnosis of bronchiectasis in medical follow up at the Pulmonary Disease Clinic of the School of Medicine of the Universidade de São Paulo. After verbal and written explanations of the study, those who agree to participate will sign a statement of informed consent approved by the Human Research Ethics Committee of Universidade Nove de Julho. The group of healthy patients will be composed of patients in treatment at the dental clinic of Universidade Nove de Julho, who will receive clarifications regarding the study and will also sign a statement of informed consent. The study will be conducted in compliance with the precepts stipulated in the Declaration of Helsinki (revised in Fortaleza, Brazil, 2013).

Calculation of sample size - To achieve an effect size of 0.40 among the four groups (PDT in healthy participants. PDT in patients with bronchiectasis, periodontal treatment or denture hygiene in healthy participants, periodontal treatment or denture hygiene in patients with bronchiectasis), assuming an alpha error of 0.05 and beta error of 0.80, the total sample will be 80 individuals (20 per group). The sample size calculation was performed using G*Power (version 3.1.9.2) (Faul, 2007).

Inclusion criteria - Men and women aged 60 years or older, with or without a diagnosis of bronchiectasis, with more than 10 natural teeth or using complete upper and lower dentures.

Exclusion criteria - smokers or ex-smokers having quit less than five years ago, a diagnosis of cystic fibrosis (which, although is a lung disease, has a genetic etiology) and hypersensitivity to the photosensitizing agent used in PDT.

Training and calibration of examiner - An examiner (gold standard) will perform training and calibration exercises to maximize the reproducibility of the measurements. For such, 10 individuals with halitosis will be evaluated using the Oral Chroma® device. These individuals will not participate in the main study. The intraclass correlation coefficient (ICC) will be calculated for the determination of intra-examiner agreement (≥ 0.90) with regard to the halitosis readings.

Randomization - The 40 healthy dentate individuals will be randomized in two groups: Group A (20 individuals submitted to treatment with a tongue scraper) and Group B (20 individuals submitted to treatment with PDT). The 40 healthy edentulous individuals will be randomized in two groups: Group C (20 individuals submitted to treatment with a tongue scraper) and Group D (20 individuals submitted to treatment with PDT). Therefore, two independent randomizations will be performed for these distinct groups of individuals (dentate and edentulous). Opaque envelopes will be identified with sequential numbers (1 to 40) and will contain pieces of paper with the information of the corresponding experimental group (A or B and C or D). Block randomization will be performed in blocks of five patients (four blocks for both treatments; example of a block: AABAB). The envelopes will be sealed and kept in numerical order in a safe place until the time of the treatments. The randomization and preparation of the envelopes will be performed by a researcher who will not otherwise participate in the study. The same procedure will be performed for the patients with bronchiectasis. Randomization will be performed using Microsoft Excel, version 2013.

Characterization of the study - The experimental design will consist of four groups: G1- healthy older adults with halitosis and 10 teeth or more (n = 40); G2- healthy older adults with halitosis who wear complete dentures (n = 40); G3- older adults with bronchiectasis who have halitosis and 10 teeth or more (n = 40); and G4- older adults with bronchiectasis who have halitosis and wear complete dentures (n = 40). The evaluation of halitosis and the microbiological analysis of the dorsum of the tongue will be performed at baseline (1st session), after treatment with PDT, periodontal treatment or denture hygiene (2nd session) and after three months (3rd session)

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years or older
* Halitosis positive: ≥ 112 ppbin the gas chromatography test
* Patients with or without a diagnosis of bronchiectasis
* Patients with more than 10 natural teeth or using complete upper and lower dentures.

Exclusion Criteria:

* Smokers or ex-smokers having quit less than five years ago
* Patients with a diagnosis of cystic fibrosis (which, although is a lung disease, has a genetic etiology)
* Patients with hypersensitivity to the photosensitizing agent used in PDT

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Halimetry (gas chromatography test) | study completion an average of 1 year
  The portable Oral ChromaTM will be used for the assessment of halitosis. A syringe will be placed in the patient's mouth with the plunger completely inserted and the participant will breathe through the nose with the mouth closed for one minute.The plunger will then be withdrawn to fill the chamber with air. This procedure will be repeated. The gas injection needle will be placed on the syringe and the plunger will be adjusted to 0.5 ml. This air will be injected into the input of the device in a single motion. This procedure will be done before and immediately after treatment.

SECONDARY OUTCOMES:
Microbiological evaluation of tongue coating | study completion an average of 1 year
  for the identification of the bacteria P. gingivalis and T. denticola.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho (UNINOVE), São Paulo, Brazil